CLINICAL TRIAL: NCT00000390
Title: Antidepressant Treatment of AIDS Related Depression.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GEIGY Pharmaceuticals (Industry)
Organization: National Institute of Mental Health (NIMH) (NIH)
Purpose: Treatment
Other Study IDs: R01MH042952 (NIH); 87-DEP (Other: GEIGY Pharmaceuticals)
Record Dates: First submitted 2000-01-17; First posted 2000-01-18 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2000-04

CONDITIONS: Depression
Keywords: Adult; Acquired Immunodeficiency Syndrome; Depression; Female; Human; Imipramine; Male; Middle Age; Acquired Immunodeficiency Syndrome -- *complications; Depression -- *drug therapy; Depression -- etiology; Imipramine -- *therapeutic use
MeSH Terms: conditions — Depression; Acquired Immunodeficiency Syndrome | interventions — Imipramine

INTERVENTIONS:
Drug: Imipramine hydrochloride

SUMMARY:
To test the effectiveness treating AIDS related depression with imipramine hydrochloride.

Depression syndromes are commonly associated with chronic, disabling, and fatal diseases. Due to the relentless course of HIV infection, there is a certain reluctance to treat the associated depression. In other illness, it has been proven that treating the depression often results in improvement of overall health status.

This is a placebo controlled trial. Half of the patients are given imipramine hydrochloride every day for 6 weeks. Assessment is done by self reports and the Hamilton Depression Rating Scale. Prior to entry all patients are given a psychiatric evaluation. There is a cross over phase in which placebo non responders are entered into an open-label study and given imipramine hydrochloride.

DETAILED DESCRIPTION:
To test the effectiveness treating AIDS related depression with imipramine hydrochloride.

Depression syndromes are commonly associated with chronic, disabling, and fatal diseases. Due to the relentless course of HIV infection, there is a certain reluctance to treat the associated depression. In other illness, it has been proven that treating the depression often results in improvement of overall health status.

This is a placebo controlled trial. Half of the patients are given imipramine hydrochloride every day for 6 weeks. Assessment is done by self reports and the Hamilton Depression Rating Scale. Prior to entry all patients are given a psychiatric evaluation. There is a cross over phase in which placebo non responders are entered into an open-label study and given imipramine hydrochloride.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ambulatory and relatively good health. Even if unable to work at least able to partially care care for self and not demented.
* May have been alcoholic or drug abuser 6 months previous.
* Unspecified
* CD4 Unspecified.

Exclusion Criteria:

* Non ambulatory patients or those requiring extensive help in self care are excluded.
* Non ambulatory patients or those requiring extensive help in self care are excluded.
* Current alcohol or drug abuse.
* Unspecified

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Frances A, Study Chair; Manning D, Study Chair
Locations (1):
- New York Hosp - Cornell Med Ctr, New York, New York, United States